CLINICAL TRIAL: NCT03138603
Title: Metoprolol to Reduce Perioperative Myocardial Injury
Acronym: ORION
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB19-1797; 5R01HL126892 (NIH)
Record Dates: First submitted 2017-04-26; First posted 2017-05-03 (Actual); Results first posted 2025-02-05 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Heart Diseases
Keywords: surgery; heart disease; metoprolol; myocardial injury; coronary artery disease
MeSH Terms: conditions — Heart Diseases; Coronary Artery Disease | interventions — Metoprolol; Adrenergic beta-Antagonists; salicylhydroxamic acid

STUDY DESIGN:
Intervention Model Description: Single-center, double blinded placebo controlled
Who Masked: Participant, Care Provider, Investigator
Masking Description: Double blind masking
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Metoprolol (Experimental): Metoprolol group, 3-intravenous doses of 5mg metoprolol tartrate (over 15-minutes), and oral dose(s) of 25mg metoprolol approximately every 8 hours postoperatively for up to 3-days (or 72 hrs).
  Interventions: Drug: Metoprolol Tartrate
- Placebo (Placebo Comparator): Placebo comparator group, up-to-three intravenous doses of placebo comparator (over 15-minutes), and oral dose(s) of a placebo comparator approximately every 8 hours postoperatively for up to 3-days (or 72 hrs).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Metoprolol Tartrate — Patients will be randomly assigned to receive up-to-three intravenous doses of 5mg metoprolol tartrate (over 15-minutes) at the end of their surgical procedure, and a scheduled oral dose regimen of 25mg metoprolol approximately every 8-hours postoperatively for up to 3-days (or 72 hrs).
  Other Names: Beta-blocker
  Arms: Metoprolol
Drug: Placebo — Patients will be randomly assigned to receive up-to-three intravenous doses of a placebo-comparator (over 15-minutes) at the end of their surgical procedure, and scheduled oral dose regimen of a placebo-comparator approximately every 8-hours postoperatively for up to 3-days (or 72 hrs).
  Other Names: Sham; Placebo-comparator; Control
  Arms: Placebo

SUMMARY:
The purpose of this research study is to test if a commonly used, FDA-approved medication, called metoprolol, given at the conclusion of anesthesia following surgery, and during postoperative admission, reduces the possibility of heart related complications in patients with coronary artery disease (CAD).

DETAILED DESCRIPTION:
All enrolled patients will be beta-blocker naïve for at least 30-days prior to their scheduled surgical procedure. Study patients will be randomly assigned to an interventional drug arm (metoprolol tartrate vs placebo-comparator). At the conclusion of anesthesia following the surgical procedure, patients hemodynamically stable and meeting study safety parameters (heart rate greater-than-65; systolic blood pressure greater-than-110) will receive 3-intravenous doses of interventional study drug (metoprolol tartrate 5mg or placebo-comparator), based on previously assigned study arm; then, patients remaining hemodynamically stable will receive an oral dose (25mg metoprolol vs placebo-comparator) approximately every 8-hours for up to 3-days during postoperative hospital admission.

From arrival in the preop holding area through up to 72 hours postoperative admission to hospital discharge or end of study treatment (whichever occurs first), patients will be continuously monitored through medical records assessments, Holter monitoring, mobile hemodynamic monitoring (VisiMobile), and in-person daily follow-up visits that include 12-lead ECG, and blood collections for serial cardiac biomarkers for high-sensitivity troponin.

Additional study patient postoperative assessment will be performed at 30 days and 1 year after surgery. These can be completed by interview and/or medical record review.

ELIGIBILITY:
Inclusion Criteria

1. Age >= 50 years
2. Beta-blocker naïve [30 days prior to surgery]
3. Previously diagnosed coronary artery disease (CAD), or

   1. History of peripheral vascular disease (PVD), or
   2. Chronic kidney disease (CKD) [eGFR ≤60ml/min], or
   3. History of positive stress test or
   4. At high risk for CAD (must meet at least 2 criteria):

   i. Age >= 70 years ii. Hypertension iii. Diabetes requiring oral medication or insulin iv. Current smoker or some days smoker within the past 2 years
4. Major non-cardiac, elective surgery under general anesthesia

Exclusion Criteria

Subjects will not be enrolled if any of the following criteria exist:

1. History of stroke, or transient ischemic attack (TIA)
2. Previously diagnosed carotid disease, i.e., either 70% unilateral or 50% bilateral carotid occlusion.
3. Heart rate <=55bpm
4. Congestive heart failure with New York Heart Association(NYHA) Functional Classification of III-IV or left ventricular heart failure with ejection fraction ≤50%
5. Severe valvular regurgitation
6. Second or third degree atrioventricular (AV) block without pacemaker
7. Active asthma or chronic obstructive pulmonary disease (COPD) with symptoms or resolving symptoms on day of surgery
8. Anemia [HB<=9g/dL]
9. Allergy to beta-blockade drugs
10. Unwilling or unable to give consent for participation
11. Undergoing any carotid endarterectomy, endovascular, endoscopic, superficial, or ambulatory procedures
12. Pregnancy or lactating women
13. Prisoners

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2023-04-18 (Actual); Study Completion 2023-08-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Nagele, MD, Principal Investigator — University of Chicago Medicine
Locations (2):
- United States (2):
  - University of Chicago Medicine, Chicago, Illinois
  - Washington University School of Medicine, St Louis, Missouri

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Metoprolol | Placebo
Started | 34 | 38
Completed | 34 | 38
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Metoprolol | Placebo | Total
Number analyzed (Participants) | 34 | 38 | 72
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 4 | 6 | 10
  >=65 years | 30 | 32 | 62
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 19 | 43
  Male | 10 | 19 | 29
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 33 | 38 | 71
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 7 | 5 | 12
  White | 26 | 30 | 56
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 34 | 38 | 72

OUTCOME MEASURES:

1. Primary Outcome: Effectiveness of Beta-blocker Therapy Reducing Post-operative Myocardial Injury
Description: Measured effectiveness of post-operative beta-blocker therapy to reduce myocardial injury by monitoring daily biomarkers (High-Sensitivity cardiac Troponin [HS-cTn]).
  Daily post-operative biomarker (hs-cTn) measurements to determine myocardial injury.
  Myocardial injury is defined as a new hscTn elevation >99th percentile, or a 50% increase if the baseline hscTn is already elevated >99th percentile
Time Frame: 0-3 days, following surgery
Population: Analysis is comprised of participants meeting criteria for randomization to receive intervention, with biomarker (hs-cTn) showing increased value(s).
Measure: Number; unit: participants
Groups:
- Metoprolol: Metoprolol group, 3-intravenous doses of 5mg metoprolol tartrate (over 15-minutes), and oral dose(s) of 25mg metoprolol approximately every 8 hours postoperatively for up to 3-days (or 72 hrs).
  Metoprolol Tartrate: Patients will be randomly assigned to receive up-to-three intravenous doses of 5mg metoprolol tartrate (over 15-minutes) at the end of their surgical procedure, and a scheduled oral dose regimen of 25mg metoprolol approximately every 8-hours postoperatively for up to 3-days (or 72 hrs).
  Post-operative analysis to determine Myocardial Injury (hs-cTnT) in randomized metoprolol group.
- Placebo: Placebo comparator group, up-to-three intravenous doses of placebo comparator (over 15-minutes), and oral dose(s) of a placebo comparator approximately every 8 hours postoperatively for up to 3-days (or 72 hrs).
  Placebo: Patients will be randomly assigned to receive up-to-three intravenous doses of a placebo-comparator (over 15-minutes) at the end of their surgical procedure, and scheduled oral dose regimen of a placebo-comparator approximately every 8-hours postoperatively for up to 3-days (or 72 hrs).
  Post-operative analysis to determine Myocardial Injury (hs-cTnT) in randomized placebo group.
Arm/Group | Metoprolol | Placebo
Number analyzed (Participants) | 34 | 38
participants | 9 | 11

2. Secondary Outcome: Effectiveness in Reduction of Major Adverse Cardiac Events (MACE)
Description: MACE are defined as myocardial ischemia (MI), cardiac death or coronary revascularization
Time Frame: 0-3 days, following surgery
Population: MACE analysis is comprised of eligible participants meeting criteria for randomization to receive intervention, having myocardial ischemia, cardiac death, or coronary revascularization.
Measure: Number; unit: participants
Arm/Group | Metoprolol | Placebo
Number analyzed (Participants) | 34 | 38
participants | 0 | 0

3. Secondary Outcome: Monitor Post-operative Myocardial Ischemia
Description: Post-operative cardiac monitoring via ECG to evaluate if myocardial ischemia is present.
  Myocardial Ischemia is defined as ST depression or elevation of ≥0.2 mV in one lead or ≥0.1 mV in two contiguous leads lasting ≥10 min
Time Frame: 0-3 days, following surgery
Population: Analysis is comprised of eligible participants meeting criteria for randomization to receive intervention, with post-operative cardiac monitoring (ECG), showing myocardial ischemia is present.
  Myocardial Ischemia is defined as ST depression or elevation of ≥0.2 mV in one lead or ≥0.1 mV in two contiguous leads lasting ≥10 min
Measure: Count of Participants; unit: Participants
Arm/Group | Metoprolol | Placebo
Number analyzed (Participants) | 34 | 38
Participants | 0 | 0

4. Secondary Outcome: Number of Stroke Related Events Following Surgery
Description: Stroke will be defined as focal or global cerebral, spinal, or retinal dysfunction of sudden onset
Time Frame: 0-3 days, following surgery
Population: Analysis is comprised of eligible participants meeting criteria for randomization to receive intervention, with post-operative sudden onset of neurological effects from cerebral dysfunction.
Measure: Count of Participants; unit: Participants
Arm/Group | Metoprolol | Placebo
Number analyzed (Participants) | 34 | 38
Participants | 0 | 0

5. Secondary Outcome: Number of Participants Having Vasopressor Therapy to Regulate Symptomatic Hypotension
Description: Monitor participants with vasopressor requirements for blood pressure regulation due to symptomatic hypotension (rate/duration time).
  Symptomatic hypotension (systolic BP < 90 mmHg) can be determined by clinical intervention due to low blood pressure and/or patient developed clinical symptoms due to hypotension.
Time Frame: 0-3 days, following surgery
Population: Analysis is comprised of eligible participants meeting criteria for randomization to receive intervention, having significant post-operative hypotension (systolic BP < 90 mmHg), requiring therapeutic intervention (vasopressor).
Measure: Count of Participants; unit: Participants
Arm/Group | Metoprolol | Placebo
Number analyzed (Participants) | 34 | 38
Participants | 0 | 0

6. Secondary Outcome: Number of Participant Incidence of Clinically Relevant Bradycardia
Description: Monitored participants with cumulative events of bradycardia (rate/duration time).
  Bradycardia is defined as low heart rate (HR < 50/min).
Time Frame: 0-3 days, following surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Metoprolol | Placebo
Number analyzed (Participants) | 34 | 38
Participants | 0 | 1

7. Secondary Outcome: Participants Number of Days Spent Post-operative Hospitalization
Description: Measurement of participants number of days spent hospitalized (0-3 days) following surgery.
Time Frame: 0-3 days following surgery
Population: Analysis is comprised of eligible participants meeting criteria for randomization to receive intervention, with post-operative length of hospital stay in days.
Measure: Median (Full Range); unit: days
Arm/Group | Metoprolol | Placebo
Number analyzed (Participants) | 34 | 38
days
  Participant post-operative hospitalization in days | 2.5 [2 to 3] | 2.5 [2 to 3]
  Participant post-operative Intensive Care Unit (ICU) hospitalization in days | 2 [2 to 3] | 3 [2 to 3]

8. Secondary Outcome: Patient Recovery Progress Events at 30-days Post-operative.
Description: Measured number of participant post-operative recovery events, 30-days following the surgical procedure.
Time Frame: 30-days from surgery
Population: Analysis is comprised of eligible participants meeting criteria for randomization to receive intervention, with post-operative 1-month follow up showing readmission since surgical discharge.
Measure: Count of Participants; unit: Participants
Arm/Group | Metoprolol | Placebo
Number analyzed (Participants) | 34 | 38
Participants | 0 | 0

9. Secondary Outcome: Participant Post-operative Mortality at 1-year Following Surgery
Description: Measured number of patient post-operative mortality at 1-year.
  Measured by 'living', 'deceased', 'date of death'.
Time Frame: 1-Year from surgery
Population: Analysis is comprised of eligible participants meeting criteria for randomization to receive intervention, deceased within 1-year of post-operative discharge.
Measure: Count of Participants; unit: Participants
Arm/Group | Metoprolol | Placebo
Number analyzed (Participants) | 34 | 38
Participants | 0 | 0

10. Other Pre Specified Outcome: Measured Number of Patient Adverse Events
Description: Number of measured participant adverse events and severity associated with low blood pressure (hypotension), low heart heart (bradycardia), nausea and vomiting; or other symptoms determined 'probably', 'possibly', 'unrelated', or 'related' to the study intervention. This includes any unplanned escalation of care admissions (e.g., Intensive Care Unit [ICU]).
  Study patient safety is monitored by the investigators (MD) with experience in critical care anesthesia, as well as an experienced clinical research team responsible for data collection and reporting of events.
Time Frame: Post-operatively, 0-3 days, and day-30
Population: Analysis is comprised of eligible participants meeting criteria for randomization to receive intervention, having post-operative adverse events.
Measure: Count of Participants; unit: Participants
Arm/Group | Metoprolol | Placebo
Number analyzed (Participants) | 34 | 38
Participants
  Hypotension | 7 | 2
  Bradycardia | 0 | 1
  Death | 0 | 0
  Cardiac Arrest | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were collected and assessed during study phase participation, e.g., intervention administration, and daily post-operative follow-up, up to 30-days post-operative.
Arm/Group | Metoprolol | Placebo
All-Cause Mortality (participants affected / at risk) | 0/34 | 0/38
Serious Adverse Events (participants affected / at risk) | 0/34 | 0/38
Other Adverse Events (participants affected / at risk) | 8/34 | 3/38
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Metoprolol (N=34) | Placebo (N=38)
MACE events (Cardiac disorders) | 0 (0) | 0 (0) — a composite of nonfatal stroke, nonfatal myocardial infarction, and cardiovascular death (e.g., Myocardial Infarction, Cardiac arrest, Stroke.)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Metoprolol (N=34) | Placebo (N=38)
Bradycardia Event (Cardiac disorders) | 0 (0) | 1 (1) — A recorded period when heart rate was below 60-beats per minute.
Hypotension event (Cardiac disorders) | 8 (8) | 2 (2) — A recorded period when systolic blood pressure reading was lower than 90 mm Hg.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-09-28): https://cdn.clinicaltrials.gov/large-docs/03/NCT03138603/Prot_SAP_000.pdf